CLINICAL TRIAL: NCT01069965
Title: Randomized, Double-blind, Placebo-controlled, Parallel Group, Multiple Dose, Multicenter Study to Assess Safety & Efficacy of BGP-15 Administered Orally 1 or 2 Times Daily With Metformin & Sulfonylurea or Metformin in T2 Diabetic Patients
Brief Title: Safety and Efficacy of BGP-15 in Patients With Type 2 Diabetes Mellitus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding support withdrawn.
Sponsor: N-Gene Research Laboratories, Inc. (Industry)
Collaborators: Integrium (Industry); Msource Medical Development GmbH (Unknown); Kinexum LLC (Unknown); Thermo Fisher Scientific, Inc (Industry); Haupt Pharma Wülfing GmbH (Unknown); Barc NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BGP-15-CLIN-IR04; 2009-013328-21 (EudraCT Number)
Record Dates: First submitted 2010-02-16; First posted 2010-02-17 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: Diabetes Mellitus
Keywords: Type 2
MeSH Terms: conditions — Diabetes Mellitus | interventions — BGP 15; BID protein, human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- 6. BGP-15 (Experimental): 400 mg BGP-15 + Placebo
  Interventions: Drug: BGP-15 400 mg QD
- 5. BGP-15 (Experimental): 200 mg BGP-15 BID
  Interventions: Drug: BGP-15 200 mg BID
- 4. BGP-15 (Experimental): 200 mg BGP-15 + Placebo
  Interventions: Drug: BGP-15 200 mg QD
- 3. BGP-15 (Experimental): Two 50 mg BGP-15 capsules by mouth in the morning; and two 50 mg BGP-15 capsules by mouth in the evening
  Interventions: Drug: BGP-15 100 mg BID
- 2. BGP-15 (Experimental): 100 mg BGP-15 + placebo
  Interventions: Drug: BGP-15 100 mg QD
- 1. Placebo (Experimental): Placebo BID
  Interventions: Drug: Placebo BID

INTERVENTIONS:
Drug: BGP-15 100 mg QD — Two 50 mg BGP-15 capsules by mouth in the morning; and two Placebo capsules by mouth in the evening
  Arms: 2. BGP-15
Drug: BGP-15 100 mg BID — One 100 mg BGP-15 capsule by mouth in the morning; and one 100 mg BGP-15 capsule by mouth in the evening
  Arms: 3. BGP-15
Drug: Placebo BID — Two Placebo capsules by mouth in the morning; and two Placebo capsules by mouth in the evening
  Arms: 1. Placebo
Drug: BGP-15 200 mg QD — Two 100 mg BGP-15 capsule by mouth in the morning; and two Placebo capsule by mouth in the evening
  Arms: 4. BGP-15
Drug: BGP-15 200 mg BID — Two 100 mg BGP-15 capsules by mouth in the morning; and two 100 mg BGP-15 capsules by mouth in the evening
  Arms: 5. BGP-15
Drug: BGP-15 400 mg QD — Two 200 mg BGP-15 capsules by mouth in the morning; and two Placebo capsules by mouth in the evening
  Arms: 6. BGP-15

SUMMARY:
This is a safety and dose finding efficacy study to evaluate the effects of BGP-15 over the dose range of 100 mg/day to 400 mg/day. Doses are applied once or twice a day for 13 weeks as add-on therapy to the combination of metformin and sulfonylurea treatment or metformin alone in patients with Type 2 Diabetes Mellitus.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, parallel group, multiple dose, multicenter study with 5 treatment arms and 1 placebo arm. Patients should be treated with both metformin and SU or metformin alone. Patients will be randomized to 100,100 + 100, 200, 200 + 200, and 400 mg/day or placebo, as an add-on to their current treatment. The study consists of 2 periods:

* A 14-day screening period for ascertaining the inclusion/exclusion criteria; and,
* A 13-week treatment period with different doses of BGP-15 or placebo as an add-on therapy to metformin and SU treatment or metformin treatment alone.

ELIGIBILITY:
Inclusion criteria

Patients meeting all of the following criteria will be eligible for enrollment:

1. Male and female patients with T2DM at time of diagnosis as defined by the American Diabetes Association (ADA) criteria;
2. Age between 30 and 70 years (inclusive);
3. HbA1c ≥7.5% - ≤12.0% at Screening, Visit 1;
4. FPG ≤270 mg/dL (15.0 mmol/L);
5. Body mass index (BMI) >27 and ≤40 kg/m2;
6. Current treatment with either metformin alone or in combination with SU. The dose of the current treatment must be stable for at least 8 weeks prior to randomization. Patients being treated with metformin must be at their optimal or near-optimal dose (≥1500 mg/day ± 500 mg/day for a range of 1000 to 2000 mg/day), and patients being treated with SU must be receiving at least one half of the maximum approved SU dose;
7. Women may be enrolled if all three of the following criteria are met:

   1. They have a negative serum pregnancy test at Screening;
   2. They are not breast feeding; and,
   3. They do not plan to become pregnant during the study AND if one of the following three criteria is met:

   i. They have had a hysterectomy or tubal ligation at least 6 months prior to signing the informed consent form; ii. They have been postmenopausal for at least 1 year; or, iii. They are of childbearing potential and will practice one of the following methods of birth control throughout the study: injectable or implantable hormonal contraception or intrauterine device; or two of the following methods of birth control throughout the study: oral or patch contraception plus a barrier contraceptive (eg, diaphragm plus spermicide, male or female condom plus spermicide, or vasectomized male partner). Abstinence, partner's use of condoms, and vasectomy are NOT acceptable methods of contraception;
8. Willingness to sign an informed consent document; and,
9. No conditions that hinder participation in the trial, as determined by the Investigator and Sponsor.

Exclusion criteria

Patients meeting any of the following criteria will be ineligible for enrollment:

1. Treatment with peroxisome proliferator-activated receptor (PPAR) agonists (including fibrates) within the last 3 months;
2. Treatment with dipeptidyl peptidase 4 (DPP-4) inhibitors, acarbose, or incretins within the last 3 months;
3. Chronic use of insulin injections within the last 1 month;
4. Hypoglycemia requiring third party assistance within the last 3 months;
5. Impaired hepatic function measured as alanine aminotransferase (ALAT) >2X the upper reference limit;
6. Impaired renal function measured as serum creatinine >150 umol/L (1.7 mg/dL);
7. Decompensated heart failure (New York Heart Association [NYHA] class III and IV);
8. Unstable angina pectoris or myocardial infarction within the last 12 months;
9. Clinically significant ECG abnormalities at screening including QTc interval (Bazett's) ≥450 msec or AV block >1st degree;
10. Uncontrolled, treated or untreated hypertension (systolic blood pressure [BP] ≥160 mmHg and/or diastolic BP ≥100 mmHg);
11. Any condition that the Investigator and/or Sponsor feel would interfere with trial participation or evaluation of the results eg, drug abuse or serious disease such as acquired immunodeficiency syndrome/human immunodeficiency syndrome (AIDS/HIV) antibodies, Hepatitis B, or Hepatitis C;
12. Pregnancy or breastfeeding, the intention to become pregnant, or judged to be using inadequate contraceptive measures;
13. History of alcohol and/or drug dependence within the last 2 years;
14. Receipt of any investigational drug or medical device within 3 months prior to this trial;
15. Fasting triglycerides >700 mg/dL at screening; or,
16. Diagnosis or treatment of cancer within the past 5 years except for excision of basal cell or squamous cell skin lesions.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2010-10; Primary Completion 2011-08 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Glycosylated Hemoglobin at Week 13 | Baseline and Week 13

SECONDARY OUTCOMES:
Change from Baseline in Fasting Plasma Glucose at Weeks 4, 8, 13 | Baseline and Weeks 4, 8, and 13
Change from Baseline in Plasma Glucose at Week 13 | Baseline and Week 13
Cardiovascular and metabolic biomarkers at Baseline and 13 weeks | Baseline and Week 13

CONTACTS AND LOCATIONS:
Overall Officials: Peter Damsbo, MD, Study Director — Kinexum LLC, Harper's Ferry, WV, USA; Robert Ratner, MD, Principal Investigator — Medstar Research Institute, Hyattsville, Maryland, USA; Ioanna Gouni-Berthold, MD, Principal Investigator — University of Cologne; Laszlo Koranyi, MD, Principal Investigator — Drug Research Center, Balatonfured, Hungary
Locations (30):
- United States (20):
  - Andrew J. Lewin Medical Corporation DBA National Research Institute, Los Angeles, California
  - Center for Clinical Trials, LLC., Paramount, California
  - Orange County Research Center, Tustin, California
  - Creekside Endocrine Associates PC, Denver, Colorado
  - Clinical Research of South Florida, Coral Gables, Florida
  - Metabolic Research Institute, Inc., West Palm Beach, Florida
  - Atlanta Pharmaceutical Research, Decatur, Georgia
  - ICCT Research International, Inc., Chicago, Illinois
  - Medstar Health Research Institute, Hyattsville, Maryland
  - The Center for Pharmaceutical Research, P.C., Kansas City, Missouri
  - Nevada Alliance Against Diabetes, Las Vegas, Nevada
  - New Hanover Medical Research, Wilmington, North Carolina
  - Piedmont Medical Research, LLC., Winston-Salem, North Carolina
  - Upstate Pharmaceutical Research, Greenville, South Carolina
  - Mountain View Clinical Research, Greer, South Carolina
  - Southeastern Research Associates, Inc., Taylors, South Carolina
  - Athens Medical Group, Athens, Tennessee
  - Juno Research, LLC., Houston, Texas
  - Juno Research, LLC., Katy, Texas
  - Cetero Research-San Antonio, San Antonio, Texas
- Germany (5):
  - Diabetespraxis Bad Mergentheim, Bad Mergentheim
  - Universitätsklinikum Köln, Cologne
  - Praxis Dr. Schätzl, Großheirath-Rossach
  - Schwerpunktpraxis Diabetes, Neuwied
  - Diabetologische Schwerpunktpraxis, Siegen
- Hungary (5):
  - DRUG Research Center Hungary Kft., Balatonfüred
  - Semmelweis University 2nd Clinic for Internal Medicine, Budapest
  - Petz Aladar Country Teaching Hospital, Dept of Diabetology and Metabolism, Győr
  - Dr. Bugyi Istvan Hospital, Diabetology Outpatient Clinic, Szentes
  - Zala County Hospital Department of Diabetology, Zalaegerszeg